CLINICAL TRIAL: NCT06824142
Title: Evaluation of the Feasibility, Practicality, and Interest of the 3D Ephemeris, a Tool for the Rehabilitation of Temporal Orientation Disorder in People With Alzheimer's Disease or Related Dementia: Monocentric Observational Pilot Study
Brief Title: Feasibility and Interest of the 3D Ephemeris for Temporal Orientation in Alzheimer's: Pilot Study
Acronym: E3D
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240896
Record Dates: First submitted 2025-02-07; First posted 2025-02-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Related dementia; Temporal disorientation; Rehabilitation; Adapted external aid
MeSH Terms: conditions — Alzheimer Disease | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluate in real-life conditions the effectiveness of an adapted external aid as a tool to support temporal orientation rehabilitation for individuals with Alzheimer's disease or related dementias in — Unlike other interventions, the E3D tool combines an intuitive, user-friendly interface with real-time temporal cues, offering a personalized experience designed to improve cognitive engagement. This external aid is aimed at fostering independence and improving daily functioning by providing clear and consistent information on time-related aspects, such as season, month, day of the week, and current date.

SUMMARY:
In geriatric care, occupational therapists use validated tools to assess abilities and performance, identifying deficiencies and proposing rehabilitation programs. Temporal orientation disorders are common, with studies showing that individuals who make mistakes in identifying time are at higher risk of dementia. Temporal orientation issues typically precede spatial orientation problems in Alzheimer's, especially in hospital settings where environmental cues are lost. Maintaining temporal orientation during hospitalization is crucial. While no effective rehabilitation tool currently exists, a new prototype has been developed to address temporal orientation disorders in Alzheimer's and dementia patients, with plans for further evaluation.

Main Objective Evaluate in real-life conditions the effectiveness of an adapted external aid, such as the Ephéméride 3D tool, in improving temporal orientation rehabilitation for individuals with Alzheimer's disease or related dementias in the mild to moderate stages.

Secondary Objectives

Assess the feasibility of establishing a routine with hospitalized patients. Gather feedback from patients, their families, and healthcare professionals regarding the external aid (usefulness, practicality, and aesthetics) as a prototype.

Evaluate the desire to continue using the tool once patients return home. Count the number of ephémérides deemed appropriate based on positive feedback from patients, families, and healthcare professionals. This figure is valuable for the company that may decide to scale up the product development. It will be calculated from the results of the attached questionnaires.

Method

This is a monocentric pilot observational study with data collection based on the following steps:

Day 5 (D5): Initial MMSE by the patient's physician. Prescription of temporal rehabilitation.

Day 6 (D6): Obtaining consent from the patient and their caregiver. Days 6 to 10 (D6 to D10): Daily assessment of the patient's knowledge of the season, year, month, day of the month (date), and day of the week without external aid (E3D).

Days 11 to 15 (D11 to D15): Daily assessment with external aid (E3D) for the same temporal knowledge.

Day 16 (D16): Interim and partial MMSE by the patient's physician. Days 17 to 21 (D17 to D21): Daily assessment without external aid (E3D). Days 22 to 26 (D22 to D26): Daily assessment with external aid (E3D). Day 27 (D27): Final and complete MMSE by the patient's physician. Days 28 to 30 (D28 to D30): Questionnaires for the patient, their caregiver, and healthcare professionals (including the study referent in the hospital).

20 patients will be included over a 1-year and 30-day period. Descriptive statistical analyses will be conducted to document patient characteristics at admission and the evolution of key parameters over time (D0 to D30). Paired statistical tests (T-tests/Chi-square) will be performed to identify significant changes between visit times. Longitudinal analyses using mixed-effects linear regression models will assess trends over time, accounting for correlations between repeated measures and evaluating differences based on the use of external aids.

Conclusion This observational study primarily aims to describe the feasibility and benefits of using the Ephéméride 3D tool to support temporal orientation rehabilitation in individuals with mild to moderate dementia.

DETAILED DESCRIPTION:
Context and Purpose In geriatric care, especially for individuals with Alzheimer's disease or other dementias, maintaining orientation in time (temporal orientation) is a critical aspect of cognitive function. Occupational therapists, using validated tools, help assess a patient's abilities and performance to identify deficiencies and propose rehabilitation programs tailored to the individual. Temporal orientation disorders, in which individuals struggle with identifying or understanding time (such as the day of the week, month, or year), are common in patients with Alzheimer's disease and related dementias. Research shows that individuals who make errors in temporal orientation-such as misidentifying the day, date, or month-are at a higher risk for developing dementia. Furthermore, temporal orientation issues often precede spatial orientation problems in Alzheimer's patients, meaning they can serve as early indicators of cognitive decline.

In hospital settings, these issues are often worsened due to the loss of personal environmental cues, which can leave patients feeling disoriented and confused. As such, maintaining temporal orientation during hospitalization is essential to reduce distress and support cognitive function. However, despite the clear importance of addressing temporal orientation in dementia care, there is currently no effective tool specifically designed to rehabilitate these deficits. This gap in care has prompted the development of a new tool, the Ephéméride 3D, a prototype external aid aimed at improving temporal orientation in individuals with mild to moderate dementia.

Main Objective The primary goal of this study is to evaluate, in real-life hospital conditions, the effectiveness of the Ephéméride 3D tool in improving temporal orientation rehabilitation for individuals with Alzheimer's disease or related dementias. Specifically, the study focuses on patients in the mild to moderate stages of the disease, where early intervention could be most beneficial.

Secondary Objectives

In addition to evaluating the tool's effectiveness, the study includes several secondary objectives:

Feasibility of Routine Establishment: The study will assess the practicality of integrating the Ephéméride 3D tool into the daily routine of hospitalized patients. This includes evaluating whether the tool can be consistently used throughout a patient's hospitalization period.

Feedback Collection: Patients, their families, and healthcare professionals will provide feedback on the usefulness, practicality, and aesthetic appeal of the Ephéméride 3D tool. This feedback will be critical for determining whether the tool meets the needs of the patients it is designed to assist.

Desire for Continued Use: The study will also investigate whether patients would be willing to continue using the tool once they are discharged from the hospital and return home. This will help gauge the long-term potential of the tool for continuous cognitive support.

Evaluation of Positive Feedback: The study will track the number of Ephémérides deemed appropriate for wider use, based on positive feedback from patients, their families, and healthcare professionals. This feedback will be used to decide whether the product should be scaled for broader development and distribution. A key metric for this evaluation will be derived from the results of questionnaires filled out by patients, their caregivers, and healthcare providers.

Methodology This study is a monocentric pilot observational study, meaning it will be conducted at a single site and will involve direct observations of patients over a defined period. The data collection process will follow a series of structured steps, including assessments of the patients' temporal knowledge at various points during the study.

Study Timeline and Procedures:

Day 5 (D5): The patient's physician will conduct an initial Mini-Mental State Examination (MMSE) to assess cognitive function and prescribe temporal orientation rehabilitation as needed.

Day 6 (D6): Consent will be obtained from both the patient and their caregiver to participate in the study.

Days 6 to 10 (D6 to D10): The patient's knowledge of time (season, year, month, day, and day of the week) will be assessed daily without the Ephéméride 3D tool, to establish a baseline for comparison.

Days 11 to 15 (D11 to D15): The patient's temporal knowledge will be assessed daily with the Ephéméride 3D tool. This period will allow the researchers to observe whether the tool has any positive impact on the patient's ability to maintain temporal orientation.

Day 16 (D16): The patient's physician will conduct an interim MMSE to measure any changes in cognitive function from the baseline.

Days 17 to 21 (D17 to D21): A second round of daily assessments will take place without the Ephéméride 3D tool to observe any reversion in the temporal orientation without external support.

Days 22 to 26 (D22 to D26): Another round of daily assessments with the Ephéméride 3D tool will take place to examine the sustained impact of the tool on temporal orientation.

Day 27 (D27): A final MMSE will be conducted to evaluate any long-term changes in cognitive function resulting from the intervention.

Days 28 to 30 (D28 to D30): Questionnaires will be completed by the patient, their caregiver, and healthcare professionals (including the study referent in the hospital) to gather their opinions on the usefulness and effectiveness of the tool.

Study Population The study will include 20 patients over the course of 1 year and 30 days, providing sufficient data for statistical analysis.

Data Analysis The analysis will involve descriptive statistics to document patient characteristics at admission and track changes over time. Statistical tests such as paired T-tests and Chi-square tests will be used to identify significant changes in temporal orientation across assessment periods. Additionally, longitudinal analyses using mixed-effects linear regression models will assess trends over time, accounting for correlations between repeated measures and evaluating the impact of the Ephéméride 3D tool on temporal orientation.

Expected Outcomes and Conclusion This observational study aims to determine whether the Ephéméride 3D tool can effectively support temporal orientation rehabilitation in individuals with Alzheimer's disease and related dementias. The study will primarily focus on the feasibility of using the tool in a hospital setting and the effectiveness of improving temporal orientation. If the tool proves successful, it could provide a practical solution for addressing temporal orientation deficits, thereby improving the overall quality of life for individuals with cognitive impairments.

The feedback gathered from patients, families, and healthcare providers will be essential in refining the tool and determining whether it is suitable for widespread use. Ultimately, the study will lay the foundation for future development and potential scaling of the Ephéméride 3D tool, with the hope of improving cognitive rehabilitation practices for individuals suffering from Alzheimer's disease and other dementias.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 65 years old.
* Patient presenting with temporal orientation impairment during the MMSE test.
* Patient with an MMSE score above 20 (mild stage) or a score between 10 and 20 (moderate stage).
* Patient who has not expressed any objection.

Exclusion Criteria:

* Presence of one or more disruptive behavioral disorders.
* Presence of confusion of unknown origin.
* Visual blindness.
* Inability to read or understand French.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: ndividuals hospitalized in a geriatric rehabilitation and follow-up care service.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Temporal Orientation Rehabilitation with the Ephéméride 3D Tool | 30 days
  This outcome measure assesses the effectiveness of the Ephéméride 3D tool in improving temporal orientation for individuals with Alzheimer's disease or related dementias in the mild to moderate stages. It is based on daily assessments of the patient's knowledge of time-related information, including season, year, month, day of the month (date), and day of the week, both with and without the use of the external aid (E3D)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Georges Clemenceau, Champcueil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS, PLEASE CONTACT SPONSOR FOR FURTHER INFORMATION